CLINICAL TRIAL: NCT04524611
Title: A Phase 3, Multicenter, Randomized, Efficacy Assessor-Blinded Study of Risankizumab Compared to Ustekinumab for the Treatment of Adult Subjects With Moderate to Severe Crohn's Disease Who Have Failed Anti-TNF Therapy
Brief Title: Study Comparing Intravenous (IV)/Subcutaneous (SC) Risankizumab to IV/SC Ustekinumab to Assess Change in Crohn's Disease Activity Index (CDAI) in Adult Participants With Moderate to Severe Crohn's Disease (CD)
Acronym: SEQUENCE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M20-259; 2020-002674-26 (EudraCT Number)
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Crohn's Disease (CD)
Keywords: Crohn's Disease (CD); Risankizumab; Ustekinumab; SKYRIZI
MeSH Terms: conditions — Crohn Disease | interventions — risankizumab; Ustekinumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Risankizumab Dose A Followed by Dose B (Experimental): Participants will receive intravenous risankizumab dose A at Week 0, 4 ,8 followed by subcutaneous (SC) risankizumab dose B every 8 weeks through Week 48. Participants who complete the Week 48 visit will continue SC risankizumab for up to an additional 220 weeks.
  Interventions: Drug: Risankizumab
- Ustekinumab (Active Comparator): Participants will receive weight-based intravenous ustekinumab at Week 0 followed by subcutaneous ustekinumab every 8 weeks through Week 48.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Risankizumab — Intravenous (IV) Infusion
  Other Names: ABBV-066; SKYRIZI
  Arms: Risankizumab Dose A Followed by Dose B
Drug: Risankizumab — Subcutaneous (SC) Injection
  Other Names: ABBV-066; SKYRIZI
  Arms: Risankizumab Dose A Followed by Dose B
Drug: Ustekinumab — Intravenous (IV) infusion
  Arms: Ustekinumab
Drug: Ustekinumab — Subcutaneous (SC) injection
  Arms: Ustekinumab

SUMMARY:
Crohn's disease (CD) is a long-lasting condition causing inflammation that can affect any part of the gut. This study will evaluate how well risankizumab works compared to ustekinumab. This study will assess change in Crohn's Disease Activity Index (CDAI).

Risankizumab is an investigational drug being developed for the treatment of Crohn's Disease (CD). Ustekinumab is an approved drug for the treatment of moderate and severe CD. Participants are randomly assigned to one of the three treatment groups. Each group receives a different treatment. There is a 1 in 2 chance that participants will be assigned to ustekinumab. Around 508 adult participants with moderate to severe CD will be enrolled in approximately 307 sites worldwide.

In Part 1, participants assigned to risankizumab will receive intravenous (IV) doses of risankizumab at Week 0, 4,8 and subcutaneous (SC) doses every 8 weeks thereafter through Week 48. Participants assigned to ustekinumab will receive intravenous (IV) dose of ustekinumab at Week 0 and subcutaneous (SC) doses every 8 weeks thereafter through Week 48. In Part 2, participants who received risankizumab in Part 1 and completed the Week 48 visit will continue to receive SC risankizumab for up to an additional 220 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Crohn's disease (CD) for at least 3 months prior to Baseline.
* Crohn's disease activity index (CDAI) score 220 - 450 at Baseline.
* Confirmed diagnosis of moderate to severe Crohn's Disease as assessed by stool frequency (SF), abdominal pain (AP) score, and Simple Endoscopic score for CD (SES-CD).
* Demonstrated intolerance or inadequate response to one or more anti-tumor necrosis factor (TNF) therapies.

Exclusion Criteria:

* Current diagnosis of ulcerative colitis or indeterminate colitis.
* Receipt of CD approved biologic agents prior to Baseline (as detailed in protocol), or any investigational biologic or other agent or procedure prior to Baseline (as detailed in protocol).
* Prior exposure to p19 and/or p40 inhibitors (e.g., risankizumab and ustekinumab).
* Currently know complications of CD (strictures, short bowel, etc).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Clinical Remission at Week 24 | Week 24
  Clinical remission is defined as Crohn's disease activity index (CDAI)<150.
Percentage of Participants Achieving Endoscopic Remission | Week 48
  Endoscopic remission is defined as Simple Endoscopic Score for Crohn's Disease (SES-CD) <= 4 and at least a 2-point reduction versus Baseline and no sub score greater than 1 in any individual variable, as scored by a central reviewer.
Number of Participants Reporting Adverse Events | Up to 220 Weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Clinical Remission at Week 48 | Week 48
  Clinical remission is defined as Crohn's disease activity index (CDAI)<150.
Percentage of Participants Achieving Endoscopic Response at Week 48 | Week 48
  Endoscopic response is defined as decrease in Simple Endoscopic Score for Crohn's Disease (SES-CD) > 50% from Baseline (or for participants with isolated ileal disease and a Baseline SES-CD of 4, at least a 2-point reduction from Baseline).
Percentage of Participants Achieving Endoscopic Response at Week 24 | Week 24
  Endoscopic response is defined as decrease in Simple Endoscopic Score for Crohn's Disease (SES-CD) > 50% from Baseline (or for participants with isolated ileal disease and a Baseline SES-CD of 4, at least a 2-point reduction from Baseline).
Percentage of Participants Achieving Steroid-Free Endoscopic Remission | Week 48
  Steroid-free endoscopic remission is defined as participants with endoscopic remission and not receiving steroids at Week 48.
Percentage of Participants Achieving Steroid-Free Clinical Remission | Week 48
  Steroid-free clinical remission is defined as participants with clinical remission and not receiving steroids at Week 48.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (300):
- United States (72):
  - Advanced Gastroenterology, P.C /ID# 224396, Chandler, Arizona
  - Southern California Res. Ctr. /ID# 223484, Coronado, California
  - Hoag Memorial Hosp Presbyterian /ID# 224373, Irvine, California
  - United Medical Doctors /ID# 223486, Los Alamitos, California
  - TLC Clinical Research Inc /ID# 223467, Los Angeles, California
  - Duplicate_UC Davis Medical Center /ID# 225700, Sacramento, California
  - Duplicate_University of California, San Francisco /ID# 223621, San Francisco, California
  - Duplicate_Western Connecticut Medical Group /ID# 223478, Danbury, Connecticut
  - Duplicate_Medical Research Center of CT /ID# 223540, Hamden, Connecticut
  - Yale Univ Digestive Diseases /ID# 224463, New Haven, Connecticut
  - Omega Research Maitland, LLC /ID# 223463, DeBary, Florida
  - Nature Coast Clinical Research - Inverness /ID# 223600, Inverness, Florida
  - University of Miami /ID# 223496, Miami, Florida
  - Gastroenterology Group Naples /ID# 223516, Naples, Florida
  - Advanced Research Institute, Inc /ID# 223470, New Port Richey, Florida
  - Endoscopic Research, Inc. /ID# 223505, Orlando, Florida
  - Duplicate_University of South Florida /ID# 224733, Tampa, Florida
  - Atlanta Gastro Assoc /ID# 223537, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, LLC /ID# 223525, Macon, Georgia
  - The University of Chicago DCAM /ID# 223520, Chicago, Illinois
  - NorthShore University-Endeavor Health Evanston Hospital /ID# 223538, Evanston, Illinois
  - Southwest Gastroenterology /ID# 223509, Oak Lawn, Illinois
  - University of Louisville Hospital /ID# 223471, Louisville, Kentucky
  - GI Alliance /ID# 223508, Baton Rouge, Louisiana
  - Nola Research Works, LLC /ID# 223489, New Orleans, Louisiana
  - Louisiana Research Center, LLC /ID# 223503, Shreveport, Louisiana
  - Duplicate_MGG Group Co, Inc.Chevy Chase Clinical Research /ID# 223499, Chevy Chase, Maryland
  - Gastro Center of Maryland /ID# 223518, Columbia, Maryland
  - Massachusetts General Hospital /Id# 224335, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center /ID# 228094, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 223597, Ann Arbor, Michigan
  - AA Medical Research Center - Flint /ID# 224384, Flint, Michigan
  - Gastroenterology Associates of Western Michigan, PLC d.b.a. West Michigan Clinic /ID# 223465, Wyoming, Michigan
  - Mayo Clinic - Rochester /ID# 223506, Rochester, Minnesota
  - Las Vegas Medical Research /ID# 223533, Las Vegas, Nevada
  - Univ New Mexico /ID# 223515, Albuquerque, New Mexico
  - NY Scientific /ID# 223479, Brooklyn, New York
  - Saratoga Schenectady Gastroenterology Associates - Burnt Hills /ID# 224048, Burnt Hills, New York
  - Intercity Advanced Gastroentertology Center /ID# 224313, Fresh Meadows, New York
  - North Shore University Hospital /ID# 224356, New Hyde Park, New York
  - The Mount Sinai Hospital /ID# 223687, New York, New York
  - Columbia Univ Medical Center /ID# 224215, New York, New York
  - Lenox Hill Hospital /ID# 223534, New York, New York
  - Univ NC Chapel Hill /ID# 224405, Chapel Hill, North Carolina
  - Duplicate_Atrium Health Wake Forest Baptist Medical Center /ID# 224406, Winston-Salem, North Carolina
  - Plains Clinical Research Center, LLC /ID# 223522, Fargo, North Dakota
  - University of Cincinnati Medical Center /ID# 224614, Cincinnati, Ohio
  - Cleveland Clinic Main Campus /ID# 223691, Cleveland, Ohio
  - DSI Research, LLC /ID# 234116, Springboro, Ohio
  - Hightower Clinical /ID# 223566, Oklahoma City, Oklahoma
  - Digestive Disease Specialists /ID# 223528, Oklahoma City, Oklahoma
  - Penn State Milton S. Hershey Medical Center /ID# 224216, Hershey, Pennsylvania
  - Guthrie Medical Group, PC /ID# 223910, Sayre, Pennsylvania
  - Digestive Disease Associates, LTD - Wyomissing /ID# 223462, Wyomissing, Pennsylvania
  - Medical University of South Carolina /ID# 223485, Charleston, South Carolina
  - Consultants in Gastroenterology - Columbia NE /ID# 224263, Columbia, South Carolina
  - Gastroenterology Associates, P.A. of Greenville /ID# 223497, Greenville, South Carolina
  - Gastro One /ID# 223539, Cordova, Tennessee
  - Vanderbilt University Medical Center /ID# 224610, Nashville, Tennessee
  - Baylor Scott & White Center for Inflammatory Bowel Diseases /ID# 223512, Dallas, Texas
  - Duplicate_DHAT Research Institute /ID# 223521, Garland, Texas
  - Vilo Research Group Inc /ID# 223513, Houston, Texas
  - Duplicate_Baylor College of Medicine - Baylor Medical Center /ID# 223488, Houston, Texas
  - Clinical Associates in Research Therapeutics of America, LLC /ID# 223510, San Antonio, Texas
  - Southern Star Research Institute, LLC /ID# 223598, San Antonio, Texas
  - Texas Digestive Disease Consultants - Southlake /ID# 224264, Southlake, Texas
  - Tyler Research Institute, LLC /ID# 223469, Tyler, Texas
  - University of Vermont Medical Center /ID# 224047, Burlington, Vermont
  - Richmond VA Medical Center /ID# 223586, Richmond, Virginia
  - Virginia Mason Hospital & Medical Center /ID# 224253, Seattle, Washington
  - Harborview Medical Center /ID# 224464, Seattle, Washington
  - West Virginia University Hospitals /ID# 223501, Morgantown, West Virginia
- Argentina (7):
  - Hospital Britanico de Buenos Aires /ID# 223432, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Hospital Italiano de Buenos Aires /ID# 224550, Ciudad Autonoma Buenos Aires, Buenos Aires F.D.
  - CINME Centro de Investigaciones Metabolicas /ID# 223447, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Gedyt /ID# 224698, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Duplicate_CEMIC /ID# 223670, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Duplicate_Sanatorio 9 de Julio /ID# 226086, San Miguel de Tucumán, Tucumán Province
  - Hospital Privado Universitario - Hospital Privado Centro Medico de Cordoba S.A. /ID# 223433, Córdoba
- Australia (5):
  - Wollongong Hospital /ID# 224688, Wollongong, New South Wales
  - Mater Misericordiae Limited /ID# 223642, South Brisbane, Queensland
  - Griffith University /ID# 223641, Southport, Queensland
  - Lyell McEwin Hospital /ID# 223643, Elizabeth Vale, South Australia
  - Monash Health - Monash Medical Centre /ID# 224599, Clayton, Victoria
- Austria (3):
  - Universitaetsklinikum St. Poelten /ID# 223437, Sankt Pölten, Lower Austria
  - Ordensklinikum Linz GmbH Barmherzige Schwestern /ID# 223440, Linz, Upper Austria
  - Medizinische Universitaet Wien /ID# 223438, Vienna, Vienna
- Belgium (11):
  - ZAS Palfijn /ID# 223907, Merksem, Antwerpen
  - Universite Libre de Bruxelles - Hopital Erasme /ID# 223902, Anderlecht, Brussels Capital
  - Cliniques Universitaires UCL Saint-Luc /ID# 223900, Brussels, Brussels Capital
  - Groupe Sante CHC - Clinique du MontLegia /ID# 223898, Liège, Liege
  - Duplicate_CHU UCL Namur - site Godinne /ID# 223905, Godinne, Namur
  - UZ Gent /ID# 223899, Ghent, Oost-Vlaanderen
  - Vitaz /Id# 224511, Sint-Niklaas, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 223901, Leuven, Vlaams-Brabant
  - AZ-Delta /ID# 223896, Roeselare, West-Vlaanderen
  - AZ Maria Middelares /ID# 223908, Ghent
  - Duplicate_CHU de Liege /ID# 223904, Liège
- Brazil (4):
  - Faculdade de Medicina do ABC /ID# 223231, Santo André, La Spezia
  - Upeclin Fmb - Unesp /Id# 223234, Botucatu, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto /ID# 223233, Ribeirão Preto, São Paulo
  - Kaiser Clinica e Hospital Dia /ID# 223232, São José do Rio Preto, São Paulo
- Bulgaria (4):
  - Hospital Tsaritsa Yoanna /ID# 223822, Sofiya, Sofia
  - Umbal Kaspela /ID# 223415, Plovdiv
  - 2nd Mhat /ID# 223425, Sofia
  - Acibadem City Clinic Tokuda University Hospital EAD /ID# 223757, Sofia
- Canada (14):
  - Duplicate_University of Calgary /ID# 223750, Calgary, Alberta
  - Allen Whey Khye Lim Professional Corporation /ID# 223755, Edmonton, Alberta
  - Covenant Health /ID# 223753, Edmonton, Alberta
  - Fraser Clinical Trials Inc /ID# 223742, New Westminster, British Columbia
  - Percuro Clinical Research, Ltd /ID# 223747, Victoria, British Columbia
  - QEII - Health Sciences Centre /ID# 223748, Halifax, Nova Scotia
  - London Health Sciences Centre - University Hospital /ID# 223741, London, Ontario
  - Scott Shulman Medicine Professional Corporation /ID# 223754, North Bay, Ontario
  - Mount Sinai Hospital /ID# 223752, Toronto, Ontario
  - Axler, Toronto, ON. Canada /ID# 223740, Toronto, Ontario
  - CISSS de la Monteregie /ID# 224399, Greenfield Park, Quebec
  - CSSS Alphonse-Desjardins, CHAU de Levis /ID# 223744, Lévis, Quebec
  - Montreal General Hospital- McGill University Health Center /ID# 223743, Montreal, Quebec
  - Duplicate_Duplicate_CHUS - Hopital Fleurimont /ID# 224819, Sherbrooke, Quebec
- Chile (3):
  - Hospital Guillermo Grant Benavente de Concepción /ID# 223668, Concepción, Bio-Bio
  - Hospital Las Higueras /ID# 223669, Talcahuano, Bio-Bio
  - Sociedad de Servicios Medicos Walsen Galmez Ltda. /ID# 224032, Providencia, Region Metropolitana Santiago
- China (21):
  - Anhui Provincial Hospital /ID# 224832, Hefei, Anhui
  - Peking University Third Hospital /ID# 224479, Beijing, Beijing Municipality
  - Chongqing General Hospital /ID# 232305, Chongqing, Chongqing Municipality
  - Zhongshan Hospital Xiamen University /ID# 224663, Xiamen, Fujian
  - Zhujiang Hospital of Southern Medical University /ID# 224524, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University /ID# 224416, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Zhengzhou University /ID# 224528, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 224545, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College of HUST /ID# 224428, Wuhan, Hubei
  - Renmin Hospital of Wuhan University /ID# 224525, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University /ID# 224684, Changsha, Hunan
  - Duplicate_The Third Xiangya Hospital of Central South University /ID# 224754, Changsha, Hunan
  - Changzhou No.2 People's Hospital /ID# 238965, Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital /ID# 224746, Nanjing, Jiangsu
  - Wuxi People's Hospital /ID# 224426, Wuxi, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 224507, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University /ID# 224478, Shenyang, Liaoning
  - Renji Hospital, Shanghai Jiaotong University School of Medicine /ID# 224420, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University /ID# 224786, Chengdu, Sichuan
  - The second affiliated hospital of Zhejiang University school of medicine /ID# 224662, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine /ID# 224421, Hangzhou, Zhejiang
- Czechia (6):
  - Iscare Klinické Centrum /ID# 223279, Prague, Praha 9
  - Nemocnice Ceske Budejovice a.s. /ID# 224219, České Budějovice
  - Hepato-Gastroenterologie HK, s.r.o. /ID# 223277, Hradec Králové
  - Nemocnice Pardubickeho kraje, a.s. /ID# 223256, Pardubice
  - Axon Clinical, s.r.o. /ID# 223260, Prague
  - Nemocnice Horovice - NH Hospital a.s /ID# 223276, Prague
- France (16):
  - Chu de Nice-Hopital L'Archet Ii /Id# 223763, Nice, Alpes-Maritimes
  - CHU Clermont-Ferrand /ID# 224529, Clermont, Auvergne-Rhône-Alpes
  - APHM - Hopital Nord /ID# 223869, Marseille, Bouches-du-Rhone
  - Duplicate_CHU Bordeaux - Hopital Haut Leveque /ID# 223764, Pessac, Gironde
  - CHU Montpellier - Hopital Saint Eloi /ID# 223860, Montpellier, Herault
  - Duplicate_CHU Grenoble - Hopital Michallon /ID# 224091, La Tronche, Isere
  - CHU Reims - Hôpital Robert Debre /ID# 224530, Reims, Marne
  - CHRU Nancy - Hopitaux de Brabois /ID# 223767, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHRU Lille - Hopital Claude Huriez /ID# 223765, Lille, Nord
  - Centre Hospitalier Universitaire de Nantes, Hotel Dieu -HME /ID# 241098, Nantes, Pays de la Loire Region
  - Centre Hospitalier Universitaire de Saint Etienne - Hopital Nord /ID# 223768, St-Priest-en-Jarez, Pays de la Loire Region
  - Clinique Jules Verne /ID# 223870, Nantes
  - Polyclinique Grand Sud /ID# 224092, Nîmes
  - Hopital Universitaire Purpan Hopital Rangueil /ID# 224732, Toulouse
  - Hopital Beaujon /ID# 223863, Clichy, Île-de-France Region
  - Centre Medico Chirurgical Ambroise Pare Hartmann /ID# 249859, Neuilly-sur-Seine, Île-de-France Region
- Germany (21):
  - Universitaetsklinikum Freiburg /ID# 223406, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitatsklinikum Mannheim /ID# 223410, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Ulm /ID# 223400, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen /ID# 223404, Erlangen, Bavaria
  - Universitatsklinik Regensburg /ID# 223407, Regensburg, Bavaria
  - Duplicate_Agaplesion Markus Krankenhaus /ID# 223673, Frankfurt am Main, Hesse
  - Universitaetsklinikum Frankfurt /ID# 223396, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover /ID# 223402, Hanover, Lower Saxony
  - Klinikum Lueneburg /ID# 223408, Lüneburg, Lower Saxony
  - Praxiszentrum fuer Gastroenterologie /ID# 223409, Grevenbroich, North Rhine-Westphalia
  - Zentrum für Gastroenterologie Saar MVZ GmbH /ID# 223482, Saarbrücken, Saarland
  - Duplicate_Universitaetsklinikum Carl Gustav Carus an der TU Dresden /ID# 223403, Dresden, Saxony
  - Eugastro /ID# 223401, Leipzig, Saxony
  - Otto-von-Guericke-Universitaet /ID# 223413, Magdeburg, Saxony-Anhalt
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 223395, Kiel, Schleswig-Holstein
  - Duplicate_Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 223405, Berlin
  - Gastroenterologische Spezialpraxis am Wittenbergplatz /ID# 229110, Berlin
  - MVZ fuer Gastroenterlogie am Bayerischen Platz /ID# 223411, Berlin
  - DRK Kliniken Berlin Westend /ID# 223412, Berlin
  - Krankenhaus Waldfriede /ID# 223397, Berlin-Zehlendorf
  - Medizinisches Versorgungszentrum Portal 10 /ID# 224552, Münster
- Greece (7):
  - General Hospital of Athens Ippokratio /ID# 223344, Athens, Attica
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 223342, Athens, Attica
  - General Hospital of Nikaia-Piraeus "Agios Panteleimon" /ID# 223340, Nikaia, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 223336, Heraklion, Crete
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 223338, Athens
  - University General Hospital of Ioannina /ID# 223339, Ioannina
  - General Hospital of Thessaloniki Hippokrateio /ID# 223887, Thessaloniki
- Hungary (5):
  - Duplicate_Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont /ID# 223774, Szeged, Csongrád megye
  - Duplicate_Debreceni Egyetem Klinikai Kozpont /ID# 223773, Debrecen, Hajdú-Bihar
  - Duplicate_Clinfan Szolgaltato Kft. /ID# 224751, Szekszárd, Tolna County
  - Clinexpert Kft /ID# 223775, Budapest
  - Semmelweis Egyetem /ID# 223772, Budapest
- Israel (7):
  - Yitzhak Shamir Medical Center /ID# 224686, Ẕerifin, Central District
  - Shaare Zedek Medical Center /ID# 223549, Jerusalem, Jerusalem
  - The Edith Wolfson Medical Center /ID# 227652, Ashkelon, Southern District
  - Soroka University Medical Center /ID# 223556, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 223557, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 223551, Tel Aviv, Tel Aviv
  - Rabin Medical Center /ID# 223558, Petah Tikva
- Italy (13):
  - Duplicate_IRCCS AOU di Bologna - Policlinico Sant'Orsola-Malpighi /ID# 223330, Bologna, Emilia-Romagna
  - Duplicate_Ospedale Policlinico San Martino /ID# 223329, Genoa, Genova
  - Duplicate_Ospedale San Raffaele IRCCS /ID# 241167, Milan, Milano
  - ASST Fatebenefratelli Sacco /ID# 223322, Milan, Milano
  - ASST Rhodense/Presidio Ospedaliero di Rho /ID# 223335, Rho, Milano
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 223332, Rome, Roma
  - Azienda Ospedaliera San Camillo Forlanini /ID# 223325, Rome, Roma
  - Duplicate_Policlinico Agostino Gemelli /ID# 223323, Rome, Roma
  - Duplicate_IRCCS Ospedale Sacro Cuore Don Calabria /ID# 223327, Negrar, Verona
  - Azienda Ospedaliera G. Brotzu /ID# 241165, Cagliari
  - Duplicate_Ospedale San Giovanni Di Dio - Cagliari /ID# 223474, Cagliari
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico /ID# 223324, Milan
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello /ID# 223333, Palermo
- Mexico (5):
  - Centro de Investigacion en Artritis y Osteoporosis S.C. /ID# 227179, Mexicali, Estado de Baja California
  - BRCR Global Mexico /ID# 223970, Guadalajara, Jalisco
  - Centro Medico Zambrano Hellion /ID# 224025, San Pedro Garza García, Nuevo León
  - Medical Care & Research SA de CV /ID# 223974, Mérida, Yucatán
  - Faicic S de Rl de Cv /Id# 226990, Veracruz
- Netherlands (4):
  - Radboud Universitair Medisch Centrum /ID# 233750, Nijmegen, Gelderland
  - Elisabeth Tweesteden Ziekenhuis /ID# 223229, Tilburg, North Brabant
  - Amsterdam UMC, locatie AMC /ID# 223228, Amsterdam, North Holland
  - Universitair Medisch Centrum Utrecht /ID# 223696, Utrecht
- Poland (3):
  - Gastromed Sp. z o.o /ID# 223705, Torun, Kuyavian-Pomeranian Voivodeship
  - Malopolskie Centrum Kliniczne /ID# 223708, Krakow, Lesser Poland Voivodeship
  - Vivamed Sp. z o.o. /ID# 223706, Warsaw, Masovian Voivodeship
- Romania (7):
  - Duplicate_Institutul Clinic Fundeni /ID# 223914, Bucharest, București
  - Duplicate_Univ Emergency Hosp Bucharest /ID# 223579, Bucharest, București
  - Sana Monitoring /Id# 223682, Bucharest
  - Spitalul Clinic Colentina /ID# 223680, Bucharest
  - Spitalul Clinic Judetean de Urgenta Targu Mures /ID# 224017, Târgu Mureş
  - Targu Mures Emergency Clinical County Hospital /ID# 223613, Târgu Mureş
  - Cabinet Particular Policlinic Algomed /ID# 223578, Timișoara
- Russia (3):
  - Immanuel Kant Baltic Federal University /ID# 224224, Kaliningrad, Kaliningrad Oblast
  - National Medical Research Center of Coloproctology n.a. A. N. Ryzhikh /ID# 224222, Moscow
  - City Clinical Hospital No. 31 /ID# 224223, Saint Petersburg
- Slovakia (4):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica /ID# 223302, Banská Bystrica, Banská Bystrica Region
  - KM Management, spol. s.r.o. /ID# 223304, Nitra, Nitra Region
  - Fakultna nemocnica s poliklinikou Nove Zamky /ID# 224580, Nové Zámky, Nitra Region
  - Duplicate_GASTRO I., s.r.o. /ID# 223303, Prešov, Presov
- South Africa (4):
  - Lenasia Clinical Trial Centre /ID# 224306, Johannesburg, Gauteng
  - Dr MJ Prins /ID# 224304, Cape Town, Western Cape
  - Private Practice Dr MN Rajabally /ID# 223805, Cape Town, Western Cape
  - Spoke Research Inc /ID# 223803, CAPE TOWN Milnerton, Western Cape
- South Korea (4):
  - Duplicate_The Catholic University of Korea, Daejeon St.Mary's Hospital /ID# 223456, Junggu, Daejeon Gwang Yeogsi
  - Duplicate_Dong-A University Hospital /ID# 223455, 서구, Gyeongsangnam-do
  - Duplicate_Kangbuk Samsung Hospital /ID# 223452, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 223453, Seoul, Seoul Teugbyeolsi
- Spain (16):
  - Hospital Arquitecto Marcide - Complejo Hospitalario Universitario de Ferrol /ID# 223356, Ferrol, A Coruna
  - Duplicate_Hospital Clínico Universitario de Santiago-CHUS /ID# 226554, Santiago de Compostela, A Coruna
  - Hospital Universitario Germans Trias i Pujol /ID# 223436, Badalona, Barcelona
  - Duplicate_Hospital Universitario de Bellvitge /ID# 225719, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Fuenlabrada /ID# 223371, Fuenlabrada, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 223319, Majadahonda, Madrid
  - Hospital Universitario Central de Asturias /ID# 223368, Oviedo, Principality of Asturias
  - Hospital General Universitario de Alicante Doctor Balmis /ID# 223552, Alicante
  - Hospital Clinic de Barcelona /ID# 223355, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 223317, Madrid
  - Hospital Clinico San Carlos /ID# 223367, Madrid
  - Hospital Universitario La Paz /ID# 223318, Madrid
  - Hospital Universitario Virgen Macarena /ID# 223315, Seville
  - Hospital Universitario Virgen del Rocio /ID# 223476, Seville
  - Hospital Clinico Universitario de Valencia /ID# 223321, Valencia
  - Hospital Universitario y Politecnico La Fe /ID# 223314, Valencia
- Sweden (4):
  - Karolinska University Hospital Solna /ID# 223423, Solna, Stockholm County
  - GHP Stockholm Gastro Center /ID# 223420, Stockholm, Stockholm County
  - Duplicate_Falu Lasarett /ID# 227222, Falun
  - Danderyds sjukhus AB /ID# 223363, Stockholm
- Switzerland (3):
  - University Hospital Basel /ID# 223711, Basel Town, Canton of Basel-City
  - Duplicate_Universitatsspital Zurich /ID# 223712, Zurich, Canton of Zurich
  - Inselspital, Universitaetsspital Bern /ID# 223590, Bern
- Turkey (Türkiye) (4):
  - Gazi Universitesi Tip Fakultes /ID# 223386, Yenimahalle, Ankara
  - Ankara Univ Medical Faculty /ID# 223388, Ankara
  - Istanbul Universitesi-Cerrahpasa Cerrahpasa Tip Fakultesi /ID# 223387, Istanbul
  - Mersin University Medical /ID# 223385, Mersin
- Ukraine (3):
  - Lviv Regional Clinical Hospital /ID# 223661, Lviv, Lviv Oblast
  - Kyiv City Clinical Hospital No.18 /ID# 223700, Kyiv
  - Medical Center of LLC DIASERVIS /ID# 224249, Zaporizhzhia
- United Kingdom (17):
  - Addenbrooke's Hospital /ID# 223648, Cambridge, Cambridgeshire
  - Royal Devon & Exeter Hospital /ID# 223644, Exeter, Devon
  - Western General Hospital - NHS Lothian /ID# 223646, Edinburgh, Edinburgh, City of
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 223651, London, Greater London
  - St Thomas' Hospital - Guy's and St Thomas' NHS Foundation Trust /ID# 223647, London, Greater London
  - St George's University Hospitals NHS Foundation Trust /ID# 223656, London, Greater London
  - University Hospital Southampton NHS Foundation Trust /ID# 224351, Southampton, Hampshire
  - East and North Hertfordshire NHS Trust /ID# 224607, Stevenage, Hertfordshire
  - Queen Elizabeth University Hospital - NHS Greater Glasgow and Clyde /ID# 223653, Glasgow, Lanarkshire
  - Duplicate_Nottingham University Hospitals NHS Trust /ID# 224179, Nottingham, Nottinghamshire
  - Oxford University Hospitals NHS Foundation Trust /ID# 223645, Oxford, Oxfordshire
  - Belfast Health and Social Care Trust /ID# 224023, Belfast
  - Calderdale and Huddersfield NHS Foundation Trust /ID# 223654, Huddersfield
  - King's College Hospital NHS Foundation Trust /ID# 223649, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 223655, Newcastle upon Tyne
  - Northern Care Alliance NHS Group /ID# 223650, Salford
  - NHS Forth Valley /ID# 224657, Stirling

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Peyrin-Biroulet L, Atreya R, Danese S, Lindsay JO, Chapman JC, Anschutz T, Huang X, Zambrano J, van Haaren S, Joshi N, Duan WR, Cross RK. Efficacy and safety of risankizumab in patients with moderately to severely active Crohn's disease: interim results from the SEQUENCE open-label extension study. J Crohns Colitis. 2025 Dec 23;19(12):jjaf213. doi: 10.1093/ecco-jcc/jjaf213. PMID 41344313
- [Derived] Hasskamp J, Meinhardt C, Timmer A. Anti-IL-12/23p40 antibodies for induction of remission in Crohn's disease. Cochrane Database Syst Rev. 2025 May 13;5(5):CD007572. doi: 10.1002/14651858.CD007572.pub4. PMID 40357993
- [Derived] Peyrin-Biroulet L, Chapman JC, Colombel JF, Caprioli F, D'Haens G, Ferrante M, Schreiber S, Atreya R, Danese S, Lindsay JO, Bossuyt P, Siegmund B, Irving PM, Panaccione R, Cao Q, Neimark E, Wallace K, Anschutz T, Kligys K, Duan WR, Pivorunas V, Huang X, Berg S, Shu L, Dubinsky M; SEQUENCE Study Group. Risankizumab versus Ustekinumab for Moderate-to-Severe Crohn's Disease. N Engl J Med. 2024 Jul 18;391(3):213-223. doi: 10.1056/NEJMoa2314585. PMID 39018531
- See also: Related Info — https://www.abbvieclinicaltrials.com/